CLINICAL TRIAL: NCT00329108
Title: A Multicenter, Randomized, Double-Blind, Parallel Group Study, Comparing The Efficacy And Tolerability Of Ziprasidone (Zeldox, Geodon) vs. Olanzapine (Zyprexa) In The Treatment And Maintenance Of Response In Patients With Acute Mania
Brief Title: Ziprasidone And Olanzapine's Outcomes In Mania
Acronym: ZOOM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Please see Brief Summary for Termination Reason.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1281147
Record Dates: First submitted 2006-05-05; First posted 2006-05-24 (Estimated); Results first posted 2009-03-13 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Acute Mania; Bipolar Disorder, Manic
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone; Olanzapine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: ziprasidone hydrochloride
- B (Active Comparator)
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: ziprasidone hydrochloride — Ziprasidone will be initiated at 80 mg/day on Day 1 and titrated to 120 mg/day from Day 3. From Day 7 the dosage may be adjusted on the basis of clinical status between 120 and 160 mg/day.
  Other Names: Geodon, Zeldox
  Arms: A
Drug: olanzapine — Olanzapine will be started at 15 mg/day on Day 1 until Day 7. The dosage will then be adjusted on the basis of clinical status between 15 and 20 mg/day.
  Arms: B

SUMMARY:
The purpose of this study is to compare the efficacy and tolerability of ziprasidone versus olanzapine in the treatment of acute mania. An open label extension will further evaluate the efficacy, safety, and tolerability of ziprasidone compared with olanzapine. Study recruitment was stopped due to difficulty in enrolling the targeted number of patients on July 30, 2007. Subjects that were enrolled at the time completed the study as per protocol. There were no safety concerns involved in the decision to stop enrollment. The Last Subject Last Visit was January 10, 2008.

ELIGIBILITY:
Inclusion Criteria:

* Have a primary diagnosis of Bipolar I Disorder, current episode manic (DSM-IV 296.4x) or mixed (DSM-IV296.6x) as determined by a structured clinical interview (Mini International Neuropsychiatric Interview (MINI)) at screening.
* A minimum score of 20 on the YMRS (Youngs Mania Rating Scale).

Exclusion Criteria:

* Have a diagnosis of learning disability or organic brain syndrome.
* Have a substance-induced psychotic disorder or behavioral disturbance thought to be due to substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-11; Primary Completion 2007-07 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- Germany (3):
  - Pfizer Investigational Site, Aachen
  - Pfizer Investigational Site, Augsburg
  - Pfizer Investigational Site, Freiburg im Breisgau
- Pfizer Investigational Site, Athens, Greece
- Italy (9):
  - Pfizer Investigational Site, S. Arsenio, Salerno
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Guardiagrele (CH)
  - Pfizer Investigational Site, Lido Di Camaiore (LU)
  - Pfizer Investigational Site, Partinico (Pa)
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Siena
  - Pfizer Investigational Site, Torino
  - Pfizer Investigational Site, Trieste
- Spain (4):
  - Pfizer Investigational Site, Terrassa, Barcelona
  - Pfizer Investigational Site, Alava, Vitoria
  - Pfizer Investigational Site, Granada
  - Pfizer Investigational Site, Málaga
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Ankara
  - Pfizer Investigational Site, Istanbul

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281147&StudyName=Ziprasidone%20And%20Olanzapine%27s%20Outcomes%20In%20Mania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 47 centers in Europe.
Pre-assignment Details: After a wash out period of at least 24 hours, patients were randomized to ziprasidone or olanzapine.
Groups:
- Ziprasidone: Ziprasidone was initiated at a dosage of 80 mg/day (40 mg BID) on Day 1 and then was titrated to 120 mg/day (60 mg BID) from Day 3. From Day 7, the dosage was adjusted between 120 to 160 mg/day on the basis of clinical status at the investigator's discretion.
- Olanzapine: Olanzapine was started at 15 mg/day (15 mg once daily [QD]) on Day 1, and remained at this dosage until Day 7. The dosage was adjusted on the basis of clinical status up to 20 mg/day at the investigator's discretion.
Period: Overall Study
Arm/Group | Ziprasidone | Olanzapine
Started | 15 (study terminated due to poor recruitment) | 14 (study terminated due to poor recruitment)
Completed | 5 | 2
Not Completed | 10 | 12
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 3 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — symptomatic deterioration | 1 | 1
Not completed — Subject no longer willing to participate | 2 | 2
Not completed — study terminated by sponsor | 1 | 0
Not completed — withdrew patient after SAE resolved | 1 | 0
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone | Olanzapine | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Customized [Number; unit: participants]
  18-44 years | 9 | 7 | 16
  45-64 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Mean Reduction in Young Mania Rating Scale (YMRS) Score During the Double Blind Phase.
Description: YMRS is 11-item instrument with scales between 0 to 4 for 7 items and scales between 0 and 8 for 4 items. 0 is normal and either 4 or 8 is the highest level of abnormal, depending on the item.
Time Frame: 4 weeks
Population: Study was terminated due to poor recruitment and no efficacy data were summarized due to very low sample size. Only safety data were summarized.
Arm/Group | Ziprasidone | Olanzapine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in Clinical Global Impressions Scale for Use in Bipolar Illness Scores; Montgomery Asberg Depression Scale Scores in the Double Blind Phase.
Time Frame: up to 10 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in Global Assessment of Functioning Scale Scores, Treatment Satisfaction Questionnaire for Medication, Quality of Life Enjoyment and Satisfaction Questionnaire in the Double Blind Phase.
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Percentage of Patients With Symptomatic Remission After 4, 6 and 10 Weeks of Treatment and at the End of the Double-blind Phase.
Time Frame: 4, 6 and 10 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Time to Symptomatic Remission in the Double Blind Phase.
Time Frame: up to 10 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Patients With Clinical Response After 6 Weeks of Double-blind Treatment.
Time Frame: 6 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Percentage of Patients With Symptomatic Relapse of Mania and/or Symptomatic Relapse of Depression During the Open Label Phase.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ziprasidone | Olanzapine
Serious Adverse Events (participants affected / at risk) | 2 | 0
Other Adverse Events (participants affected / at risk) | 7 | 12
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Ziprasidone | Olanzapine
Oculogyric crisis (Eye disorders) | 1/15 | 0/14
Disease progression (General disorders) | 1/15 | 0/14
laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1/15 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Ziprasidone | Olanzapine
Anemia (Blood and lymphatic system disorders) | 0/15 | 1/14
Hyperprolactinaemia (Endocrine disorders) | 0/15 | 1/14
Dry mouth (Gastrointestinal disorders) | 0/15 | 2/14
flatulence (Gastrointestinal disorders) | 0/15 | 1/14
gingivitis (Gastrointestinal disorders) | 0/15 | 1/14
nausea (Gastrointestinal disorders) | 1/15 | 1/14
vomiting (Gastrointestinal disorders) | 1/15 | 1/14
fatigue (General disorders) | 0/15 | 2/14
pyrexia (General disorders) | 0/15 | 1/14
hypersensitivity (Immune system disorders) | 0/15 | 1/14
nasopharyngitis (Infections and infestations) | 0/15 | 1/14
pneumonia bacterial (Infections and infestations) | 0/15 | 1/14
tonsillitis (Infections and infestations) | 0/15 | 1/14
joint dislocation (Injury, poisoning and procedural complications) | 0/15 | 1/14
weight increased (Investigations) | 1/15 | 1/14
fluid retention (Metabolism and nutrition disorders) | 0/15 | 1/14
hyperlipidaemia (Metabolism and nutrition disorders) | 0/15 | 1/14
increased appetite (Metabolism and nutrition disorders) | 0/15 | 2/14
headache (Nervous system disorders) | 1/15 | 1/14
hypotonia (Nervous system disorders) | 0/15 | 1/14
somnolence (Nervous system disorders) | 3/15 | 1/14
tremor (Nervous system disorders) | 1/15 | 3/14
anxiety (Psychiatric disorders) | 1/15 | 1/14
binge eating (Psychiatric disorders) | 0/15 | 1/14
delusion (Psychiatric disorders) | 0/15 | 1/14
depressed mood (Psychiatric disorders) | 1/15 | 0/14
depression (Psychiatric disorders) | 0/15 | 1/14
insomnia (Psychiatric disorders) | 2/15 | 0/14
mania (Psychiatric disorders) | 1/15 | 0/14
breast enlargement (Reproductive system and breast disorders) | 0/15 | 1/14
sexual dysfunction (Reproductive system and breast disorders) | 0/15 | 1/14
eczema (Skin and subcutaneous tissue disorders) | 0/15 | 1/14
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0/15 | 1/14
tooth extraction (Surgical and medical procedures) | 0/15 | 1/14

LIMITATIONS AND CAVEATS:
The study was terminated due to poor recruitment. No efficacy data were summarized due to very low sample size. Only safety data were summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.